CLINICAL TRIAL: NCT06777134
Title: Relationship Between Pelvic Floor Dysfunctions and Core Endurance, Hip Rotation Muscle Strength, Tibialis Anterior and Tibialis Posterior Muscle Activation in Patients With Multiple Sclerosis
Brief Title: Relationship Between Pelvic Floor Dysfunctions and Lower Limb Strength and Activation in MS Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Berivan Beril Kılıç (Other)
Responsible Party: Sponsor-Investigator, Berivan Beril Kılıç, Assistant Professor, Biruni University
Organization: Biruni University (Other)
Other Study IDs: 05-14
Record Dates: First submitted 2025-01-04; First posted 2025-01-15 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis; Pelvic Floor Dysfunction
Keywords: pelvic floor; multiple sclerosis; core endurance; tibialis anterior; tibialis posterior; electromyography
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with multiple sclerosis
  Interventions: Other: Assessment of pelvic floor dysfunction; Other: The Quality of Life Assessment; Other: Core endurance assessment; Other: Hip strength assessment; Other: Tibialis posterior muscle activation; Other: Tibialis anterior muscle activation

INTERVENTIONS:
Other: Assessment of pelvic floor dysfunction — Pelvic floor dysfunctions in patients with multiple sclerosis will be assessed using the Pelvic Floor Distress Inventory-20 (PFDI-20). The scale is designed to assess all symptoms related to pelvic floor disorders and the severity of the distress they cause. The PFDI-20 consists of 3 subscales and 20 items, with each item rated on a scale from 0 (none) to 4 (quite a bit). To determine the scale scores, the average of the responses for each item in the subscales is multiplied by 25, resulting in a subscale score ranging from 0 to 100, and a total score ranging from 0 to 300. The Turkish validity and reliability of the scale were conducted by Çelenay et al.
Other: The Quality of Life Assessment — The quality of life of the patients will be assessed using the Multiple Sclerosis International Quality of Life Questionnaire. The questionnaire consists of 31 questions and 9 subscales. The lowest score that can be obtained from the scale is 0, the highest score is 124, and a high score indicates a low quality of life. The subscales of the questionnaire include daily living activities, psychological well-being, relationships with friends, symptoms, relationships with family, relationships with the healthcare system, emotional and sexual life, coping, and rejection. The Turkish validation of the questionnaire has been conducted.
Other: Core endurance assessment — Core endurance in patients will be assessed using McGill's core endurance tests Trunk Flexor Test: Patients sit at a 60° trunk angle with knees bent, arms crossed, and feet stabilized. Time holding the position is recorded.
  Trunk Extensor Test: Patients lie prone with the pelvis stabilized, lift the upper body above table level, and hold. Time is recorded until the body drops.
  Lateral Trunk Test: In a modified side plank (knees bent, elbow support), patients lift hips off the mat. Time is recorded until hips lower or extra support is needed.
Other: Hip strength assessment — The assessment of hip strength will specifically focus on the hip adductor and hip external rotator muscle strength. Both muscle groups are considered to be associated with the pelvic floor. Among the hip external rotators, the piriformis muscle functions as an internal stabilizer for the hip joint, while the obturator internus muscle shares fascial connections with the pelvic floor, playing a significant role in pelvic floor function. MR and EMG studies have demonstrated that the levator ani and gluteus maximus muscles are morphologically and functionally connected, and that the contraction of hip adductor and gluteal muscles facilitates the synergistic contraction of pelvic floor muscles. Based on this information, a handheld dynamometer will be used to measure the strength of the two muscle groups planned for evaluation. Measurements will be performed three times, and the average value will be recorded.
Other: Tibialis posterior muscle activation — The NeuroTrac Myoplus Pro (Quintet, Bergen, Norway) EMG device will be used for the superficial EMG analysis of the posterior tibialis muscle. During the assessment, single-use 30 x 30 mm round adhesive electrodes will be placed on the reference points. The active electrode will be positioned at the exact midpoint between the tibial tuberosity and the medial malleolus (32,33); the passive electrode will be placed 4 cm distal; and the reference electrode will be placed on the lateral malleolus.
  The patient will be asked to perform isometric plantar flexion + inversion movement of the ankle against resistance for 10 seconds. The ankle isometric contractions will be performed in 3 repetitions, with a 20-second rest period between contractions. As a result of the assessment, parameters related to the muscle's strength, total work, and resting tone will be recorded in microvolts; the maximal voluntary contraction will be recorded as a percentage.
Other: Tibialis anterior muscle activation — The NeuroTrac Myoplus Pro (Quintet, Bergen, Norway) EMG device will be used for the superficial EMG analysis of the tibialis anterior muscle. During the assessment, single-use 30 x 30 mm round adhesive electrodes will be placed on the reference points. The active electrode will be positioned on the muscle body of the tibialis anterior, the passive electrode will be placed 4 cm distal, and the reference electrode will be placed on the lateral malleolus (34,35).
  The patient will be asked to perform isometric ankle dorsiflexion against resistance for 10 seconds. The ankle isometric contractions will be performed in 3 repetitions, with a 20-second rest period between contractions. As a result of the assessment, parameters related to the muscle's strength, total work, and resting tone will be recorded in microvolts; the maximal voluntary contraction will be recorded as a percentage.

SUMMARY:
we aim to investigate the relationship between pelvic floor dysfunctions, core endurance, hip external rotation muscle strength, and tibialis posterior and tibialis anterior muscle activation in patients diagnosed with MS

ELIGIBILITY:
Inclusion Criteria:

* EDSS score between 0 and 4.0
* Having access to the internet via a high-speed smartphone or computer
* Scoring at least 21 points on the MoCA
* Having a score of Stage 3 or higher on the Functional Ambulation Scale.

Exclusion Criteria:

* Having hearing or vision problems.
* Participating in any exercise program.
* Having accompanying other neurological, cardiovascular, or orthopedic disorders.
* A history of an MS relapse or medication change within the last 6 months.
* Being in a physical condition that prevents participation in exercises.
* Comorbid conditions that negatively affect oxygen transport (e.g., severe anemia, peripheral artery disease, etc.)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is planned to include 73 patients who applied to Bakırköy Prof. Dr. Mazhar Osman Mental and Nervous Diseases Training and Research Hospital Neurology Clinic and who were diagnosed with definite Multiple Sclerosis according to McDonald Diagnostic Criteria with EDSS level between 0-4.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Pelvic floor muscle dysfunction | baseline
  Pelvic floor dysfunctions in patients with multiple sclerosis will be assessed using the Pelvic Floor Distress Inventory-20. The scale is designed to assess all symptoms related to pelvic floor disorders and the severity of the distress they cause. It consists of 3 subscales and 20 items, with each item rated on a scale from 0 (none) to 4 (quite a bit). To determine the scale scores, the average of the responses for each item in the subscales is multiplied by 25, resulting in a subscale score ranging from 0 to 100, and a total score ranging from 0 to 300. The Turkish validity and reliability of the scale were conducted.

SECONDARY OUTCOMES:
Qualitf of life | Baseline
  The quality of life of the patients will be assessed using the Multiple Sclerosis International Quality of Life Questionnaire. The questionnaire consists of 31 questions and 9 subscales. The subscales of the questionnaire include daily living activities, psychological well-being, relationships with friends, symptoms, relationships with family, relationships with the healthcare system, emotional and sexual life, coping, and rejection. An increase in the total score obtained from the scale indicates better quality of life. The Turkish validation of the questionnaire has been conducted.
Core endurance -trunk flexor endurance | baseline
  Core endurance will be assessed using McGill's tests:
  Trunk Flexor Test: Patients sit at a 60° trunk angle with knees bent, arms crossed, and feet stabilized. Time holding the position is recorded.
Core endurance -trunk extansor endurance | baseline
  Core endurance will be assessed using McGill's tests:
  Trunk Extensor Test: Patients lie prone with the pelvis stabilized, lift the upper body above table level, and hold. Time is recorded until the body drops.
Core endurance - lateral flexor endurance | baseline
  Core endurance will be assessed using McGill's tests:
  Lateral Trunk Test: In a modified side plank (knees bent, elbow support), patients lift hips off the mat. Time is recorded until hips lower or extra support is needed.
Hip strength | baseline
  The assessment of hip strength will specifically focus on the hip adductor and hip external rotator muscle strength. Both muscle groups are considered to be associated with the pelvic floor. Among the hip external rotators, the piriformis muscle functions as an internal stabilizer for the hip joint, while the obturator internus muscle shares fascial connections with the pelvic floor, playing a significant role in pelvic floor function. MR and EMG studies have demonstrated that the levator ani and gluteus maximus muscles are morphologically and functionally connected, and that the contraction of hip adductor and gluteal muscles facilitates the synergistic contraction of pelvic floor muscles. Based on this information, a handheld dynamometer will be used to measure the strength of the two muscle groups planned for evaluation. Measurements will be performed three times, and the average value will be recorded.
tibialis posterior muscle activation - peak torque | baseline
  The NeuroTrac Myoplus Pro (Quintet, Bergen, Norway) electromyography (EMG) device will be used for the superficial EMG analysis of the posterior tibialis muscle. During the assessment, single-use 30 x 30 mm round adhesive electrodes will be placed on the reference points. The active electrode will be positioned at the exact midpoint between the tibial tuberosity and the medial malleolus; the passive electrode will be placed 4 cm distal; and the reference electrode will be placed on the lateral malleolus.
  The patient will be asked to perform isometric plantar flexion + inversion movement of the ankle against resistance for 10 seconds. The ankle isometric contractions will be performed in 3 repetitions, with a 20-second rest period between contractions. As a result of the assessment, peak torque will be recorded in microvolts.
tibialis posterior muscle activation - work avarage | baseline
  The NeuroTrac Myoplus Pro (Quintet, Bergen, Norway) electromyography (EMG) device will be used for the superficial EMG analysis of the posterior tibialis muscle. During the assessment, single-use 30 x 30 mm round adhesive electrodes will be placed on the reference points. The active electrode will be positioned at the exact midpoint between the tibial tuberosity and the medial malleolus; the passive electrode will be placed 4 cm distal; and the reference electrode will be placed on the lateral malleolus.
  The patient will be asked to perform isometric plantar flexion + inversion movement of the ankle against resistance for 10 seconds. The ankle isometric contractions will be performed in 3 repetitions, with a 20-second rest period between contractions. As a result of the assessment, work avarage will be recorded in microvolts.
tibialis posterior muscle activation - percentage of maximal voluntary contractions | baseline
  The NeuroTrac Myoplus Pro (Quintet, Bergen, Norway) electromyography (EMG) device will be used for the superficial EMG analysis of the posterior tibialis muscle. During the assessment, single-use 30 x 30 mm round adhesive electrodes will be placed on the reference points. The active electrode will be positioned at the exact midpoint between the tibial tuberosity and the medial malleolus; the passive electrode will be placed 4 cm distal; and the reference electrode will be placed on the lateral malleolus.
  The patient will be asked to perform isometric plantar flexion + inversion movement of the ankle against resistance for 10 seconds. The ankle isometric contractions will be performed in 3 repetitions, with a 20-second rest period between contractions. As a result of the assessment, maximal voluntary contractions will be recorded in percentage
tibialis posterior muscle activation - rest tone | baseline
  The NeuroTrac Myoplus Pro (Quintet, Bergen, Norway) electromyography (EMG) device will be used for the superficial EMG analysis of the posterior tibialis muscle. During the assessment, single-use 30 x 30 mm round adhesive electrodes will be placed on the reference points. The active electrode will be positioned at the exact midpoint between the tibial tuberosity and the medial malleolus; the passive electrode will be placed 4 cm distal; and the reference electrode will be placed on the lateral malleolus.
  The patient will be asked to perform isometric plantar flexion + inversion movement of the ankle against resistance for 10 seconds. The ankle isometric contractions will be performed in 3 repetitions, with a 20-second rest period between contractions. As a result of the assessment, rest tone will be recorded in microvolts.
tibialis anterior muscle activation - peak torque | baseline
  The NeuroTrac Myoplus Pro (Quintet, Bergen, Norway) electromyography (EMG) device will be used for the superficial EMG analysis of the tibialis anterior muscle. During the assessment, single-use 30 x 30 mm round adhesive electrodes will be placed on the reference points. The active electrode will be positioned on the muscle body of the tibialis anterior, the passive electrode will be placed 4 cm distal, and the reference electrode will be placed on the lateral malleolus.
  The patient will be asked to perform isometric ankle dorsiflexion against resistance for 10 seconds. The ankle isometric contractions will be performed in 3 repetitions, with a 20-second rest period between contractions. As a result of the assessment, peak torque will be recorded in microvolts.
tibialis anterior muscle activation - work avarage | baseline
  The NeuroTrac Myoplus Pro (Quintet, Bergen, Norway) electromyography (EMG) device will be used for the superficial EMG analysis of the tibialis anterior muscle. During the assessment, single-use 30 x 30 mm round adhesive electrodes will be placed on the reference points. The active electrode will be positioned on the muscle body of the tibialis anterior, the passive electrode will be placed 4 cm distal, and the reference electrode will be placed on the lateral malleolus.
  The patient will be asked to perform isometric ankle dorsiflexion against resistance for 10 seconds. The ankle isometric contractions will be performed in 3 repetitions, with a 20-second rest period between contractions. As a result of the assessment, work average will be recorded in microvolts.
tibialis anterior muscle activation - percentage of maximal voluntarily contractions | baseline
  The NeuroTrac Myoplus Pro (Quintet, Bergen, Norway) electromyography (EMG) device will be used for the superficial EMG analysis of the tibialis anterior muscle. During the assessment, single-use 30 x 30 mm round adhesive electrodes will be placed on the reference points. The active electrode will be positioned on the muscle body of the tibialis anterior, the passive electrode will be placed 4 cm distal, and the reference electrode will be placed on the lateral malleolus.
  The patient will be asked to perform isometric ankle dorsiflexion against resistance for 10 seconds. The ankle isometric contractions will be performed in 3 repetitions, with a 20-second rest period between contractions. As a result of the assessment, maximal voluntary contractions will be recorded in percentage.
tibialis anterior muscle activation - rest tone | baseline
  The NeuroTrac Myoplus Pro (Quintet, Bergen, Norway) electromyography (EMG) device will be used for the superficial EMG analysis of the tibialis anterior muscle. During the assessment, single-use 30 x 30 mm round adhesive electrodes will be placed on the reference points. The active electrode will be positioned on the muscle body of the tibialis anterior, the passive electrode will be placed 4 cm distal, and the reference electrode will be placed on the lateral malleolus.
  The patient will be asked to perform isometric ankle dorsiflexion against resistance for 10 seconds. The ankle isometric contractions will be performed in 3 repetitions, with a 20-second rest period between contractions. As a result of the assessment, rest tone will be recorded in microvolts.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] İstek, A. (2009) Kronik Pelvik Ağrı Şikayeti Olan Hastalarda Posterior Tibial Sinir Uyarısı Tedavisinin (Nöromodülasyon) Yaşam Kalitesi Üzerine Etkisi
- [Result] İri, S.G. (2022) Üriner İnkontinansı Olan Kadınlarda Pelvik Taban Sağlığı Eğitimi Ve Egzersiz Programının Etkinliğinin Araştırılması
- [Result] İpeker Karagöz, F. (2022) Kadınlarda Stres Üriner İnkontinans Şiddetinin İnsülin Benzeri Büyüme Faktörü-1 Ve Kor Stabilizasyonu Üzerine Etkisinin İncelenmesi
- [Result] YAVAŞ, İpek, Özge ERTEKİN, and Turhan KAHRAMAN. "Multipl Sklerozlu Bireylerde Üriner Semptomlar, Bağırsak Semptomları ve Cinsel İşlev Bozukluğunun Tedavisinde Pelvik Taban Kas Eğitimi: Geleneksel Derleme." Turkiye Klinikleri Journal of Health Sciences/Türkiye Klinikleri Sağlık Bilimleri Dergisi 9.2 (2024).
- [Result] Yavaş, İ. (2021). Multipl sklerozlu bireylerde telerehabilitasyon temelli pelvik taban kas eğitiminin üriner inkontinans, cinsel işlev bozukluğu ve yaşam kalitesi üzerine etkisi
- [Result] Yıldız, H.C. (2018). Multipl Skleroz bireylerinde, mesane fonksiyonlarının etkilenim şiddetine göre yorgunluk, düşme, yaşam kalitesi ve pelvik taban kas kuvvetinin karşılaştırması
- [Result] Multipl sklerozun kadın cinselliği üzerine etkileri: Kontrollü çalışma Gumus H, Akpınar Z, Yılmaz H. The Journal of Sexual Medicine 11(2) 2014 p:481-485
- [Result] Nuri YILDIRIM, Niyazi AŞKAR (2017) Chronic Pelvic Floor Dysfunction Kadın Hastalıkları ve Doğum AD, Ege Üniversitesi Tıp Fakültesi, İzmir Turkiye Klinikleri J Gynecol Obst-Special Topics. 2017;10(2):210-4. https://www.turkiyeklinikleri.com/
- [Result] Chaudhry SR, Nahian A, Chaudhry K. Anatomy, Abdomen and Pelvis, Pelvis. 2023 Jul 25. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK482258/ PMID 29489173
- [Result] 10.2174/1874943701003010110
- [Result] Murley GS, Buldt AK, Trump PJ, Wickham JB. Tibialis posterior EMG activity during barefoot walking in people with neutral foot posture. J Electromyogr Kinesiol. 2009 Apr;19(2):e69-77. doi: 10.1016/j.jelekin.2007.10.002. Epub 2007 Nov 28. PMID 18053742
- [Result] Semple R, Murley GS, Woodburn J, Turner DE. Tibialis posterior in health and disease: a review of structure and function with specific reference to electromyographic studies. J Foot Ankle Res. 2009 Aug 19;2:24. doi: 10.1186/1757-1146-2-24. PMID 19691828
- [Result] Bo K, Stien R. Needle EMG registration of striated urethral wall and pelvic floor muscle activity patterns during cough, Valsalva, abdominal, hip adductor, and gluteal muscle contractions in nulliparous healthy females. Neurourol Urodyn. 1994;13(1):35-41. doi: 10.1002/nau.1930130106. PMID 8156073
- [Result] McGill SM, Childs A, Liebenson C. Endurance times for low back stabilization exercises: clinical targets for testing and training from a normal database. Arch Phys Med Rehabil. 1999 Aug;80(8):941-4. doi: 10.1016/s0003-9993(99)90087-4. PMID 10453772
- [Result] Simeoni M, Auquier P, Fernandez O, Flachenecker P, Stecchi S, Constantinescu C, Idiman E, Boyko A, Beiske A, Vollmer T, Triantafyllou N, O'Connor P, Barak Y, Biermann L, Cristiano E, Atweh S, Patrick D, Robitail S, Ammoury N, Beresniak A, Pelletier J; MusiQol study group. Validation of the Multiple Sclerosis International Quality of Life questionnaire. Mult Scler. 2008 Mar;14(2):219-30. doi: 10.1177/1352458507080733. Epub 2007 Oct 17. PMID 17942521
- [Result] Toprak Celenay S, Akbayrak T, Kaya S, Ekici G, Beksac S. Validity and reliability of the Turkish version of the Pelvic Floor Distress Inventory-20. Int Urogynecol J. 2012 Aug;23(8):1123-7. doi: 10.1007/s00192-012-1729-8. Epub 2012 Mar 29. PMID 22456806
- [Result] Afshari P, Abedi P, Majdinasab N, Tafakh S, Haghighizadeh M. Strengths of pelvic floor muscles in women with multiple sclerosis and its relationship with urinary incontinence and quality of life. Front Neurol. 2025 Jan 13;15:1514157. doi: 10.3389/fneur.2024.1514157. eCollection 2024. PMID 39871990
- [Result] Litwiller SE, Frohman EM, Zimmern PE. Multiple sclerosis and the urologist. J Urol. 1999 Mar;161(3):743-57. PMID 10022678
- [Result] Oh J, Vidal-Jordana A, Montalban X. Multiple sclerosis: clinical aspects. Curr Opin Neurol. 2018 Dec;31(6):752-759. doi: 10.1097/WCO.0000000000000622. PMID 30300239
- [Result] Sivakumar R, Jena S. Effect of unstable surface sitting on paretic anterior tibial muscle following stroke. J Bodyw Mov Ther. 2020 Jan;24(1):269-273. doi: 10.1016/j.jbmt.2019.06.001. Epub 2019 Jun 4. PMID 31987556
- [Result] Marques SAA, Silveira SRBD, Passaro AC, Haddad JM, Baracat EC, Ferreira EAG. Effect of Pelvic Floor and Hip Muscle Strengthening in the Treatment of Stress Urinary Incontinence: A Randomized Clinical Trial. J Manipulative Physiol Ther. 2020 Mar-Apr;43(3):247-256. doi: 10.1016/j.jmpt.2019.01.007. Epub 2020 Jul 21. PMID 32703614
- [Result] Wang Z, Zhu Y, Han D, Huang Q, Maruyama H, Onoda K. Effect of hip external rotator muscle contraction on pelvic floor muscle function and the piriformis. Int Urogynecol J. 2022 Oct;33(10):2833-2839. doi: 10.1007/s00192-021-05046-9. Epub 2021 Nov 29. PMID 34842941
- [Result] Barber MD, Kuchibhatla MN, Pieper CF, Bump RC. Psychometric evaluation of 2 comprehensive condition-specific quality of life instruments for women with pelvic floor disorders. Am J Obstet Gynecol. 2001 Dec;185(6):1388-95. doi: 10.1067/mob.2001.118659. PMID 11744914
- [Result] Burton C, Sajja A, Latthe PM. Effectiveness of percutaneous posterior tibial nerve stimulation for overactive bladder: a systematic review and meta-analysis. Neurourol Urodyn. 2012 Nov;31(8):1206-16. doi: 10.1002/nau.22251. Epub 2012 May 11. PMID 22581511
- [Result] Nipa SI, Sriboonreung T, Paungmali A, Phongnarisorn C. The Effects of Pelvic Floor Muscle Exercise Combined with Core Stability Exercise on Women with Stress Urinary Incontinence following the Treatment of Nonspecific Chronic Low Back Pain. Adv Urol. 2022 Sep 5;2022:2051374. doi: 10.1155/2022/2051374. eCollection 2022. PMID 36105867
- [Result] Eickmeyer SM. Anatomy and Physiology of the Pelvic Floor. Phys Med Rehabil Clin N Am. 2017 Aug;28(3):455-460. doi: 10.1016/j.pmr.2017.03.003. Epub 2017 May 27. PMID 28676358
- [Result] Bordoni B, Sugumar K, Leslie SW. Anatomy, Abdomen and Pelvis, Pelvic Floor. 2023 Jul 17. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK482200/ PMID 29489277
- [Result] Lucio AC, Perissinoto MC, Natalin RA, Prudente A, Damasceno BP, D'ancona CA. A comparative study of pelvic floor muscle training in women with multiple sclerosis: its impact on lower urinary tract symptoms and quality of life. Clinics (Sao Paulo). 2011;66(9):1563-8. doi: 10.1590/s1807-59322011000900010. PMID 22179160
- [Result] Johns JS, Krogh K, Ethans K, Chi J, Queree M, Eng JJ, Spinal Cord Injury Research Evidence Team. Pharmacological Management of Neurogenic Bowel Dysfunction after Spinal Cord Injury and Multiple Sclerosis: A Systematic Review and Clinical Implications. J Clin Med. 2021 Feb 22;10(4):882. doi: 10.3390/jcm10040882. PMID 33671492
- [Result] Miget G, Tan E, Pericolini M, Chesnel C, Haddad R, Turmel N, Amarenco G, Hentzen C. The Neurogenic Bowel Dysfunction score (NBD) is not suitable for patients with multiple sclerosis. Spinal Cord. 2022 Dec;60(12):1130-1135. doi: 10.1038/s41393-022-00837-3. Epub 2022 Jul 20. PMID 35859189
- [Result] Aguilar-Zafra S, Del Corral T, Vidal-Quevedo C, Rodriguez-Duran P, Lopez-de-Uralde-Villanueva I. Pelvic floor dysfunction negatively impacts general functional performance in patients with multiple sclerosis. Neurourol Urodyn. 2020 Mar;39(3):978-986. doi: 10.1002/nau.24314. Epub 2020 Feb 10. PMID 32040860
- [Result] Oppenheimer DR. The cervical cord in multiple sclerosis. Neuropathol Appl Neurobiol. 1978 Mar-Apr;4(2):151-62. doi: 10.1111/j.1365-2990.1978.tb00555.x. PMID 683462
- [Result] Compston A, Coles A. Multiple sclerosis. Lancet. 2008 Oct 25;372(9648):1502-17. doi: 10.1016/S0140-6736(08)61620-7. PMID 18970977
- [Result] Tullman MJ. Overview of the epidemiology, diagnosis, and disease progression associated with multiple sclerosis. Am J Manag Care. 2013 Feb;19(2 Suppl):S15-20. PMID 23544716